CLINICAL TRIAL: NCT06992661
Title: A Study of the Pharmacokinetics and Safety of Single-dose Inhaled RJ026 in Healthy Volunteers and Patients With Interstitial Lung Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jieming QU, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20250508
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Interstitial Lung Disease (ILD); Healthy Volunteers
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Experimental 1-ICD (Experimental): RJ026 inhaled powder, 4 mg, inhalation
  Interventions: Drug: RJ026 inhaled powder
- Experimental 2-ICD (Experimental): RJ026 inhaled powder, 8 mg, inhalation
  Interventions: Drug: RJ026 inhaled powder
- Experimental 3-ICD (Experimental): RJ026 inhaled powder, 12 mg, inhalation
  Interventions: Drug: RJ026 inhaled powder
- Active Comparator-ICD (Active Comparator): RJ026 600mg, Oral
  Interventions: Drug: Oral RJ026 capsules
- Experimental 1-Healthy volunteer (Experimental): RJ026 inhaled powder, 4 mg, inhalation
  Interventions: Drug: RJ026 inhaled powder
- Experimental 2-Healthy volunteer (Experimental): RJ026 inhaled powder, 8 mg, inhalation
  Interventions: Drug: RJ026 inhaled powder
- Experimental 3-Healthy volunteer (Experimental): RJ026 inhaled powder, 12 mg, inhalation
  Interventions: Drug: RJ026 inhaled powder
- Active Comparator-Healthy volunteer (Experimental): RJ026 600mg, Oral
  Interventions: Drug: Oral RJ026 capsules

INTERVENTIONS:
Drug: RJ026 inhaled powder — Developed for targeted pulmonary delivery, RJ026 utilizes a proprietary RS01 dry powder inhaler device to achieve localized therapeutic effects in lung tissue while minimizing systemic exposure.
  Preclinical studies demonstrate that inhaled administration achieves 10-20× higher lung concentrations compared to oral dosing, with correspondingly lower plasma levels - potentially reducing the hepatotoxicity risk associated with high oral doses.
  Arms: Experimental 1-Healthy volunteer; Experimental 1-ICD; Experimental 2-Healthy volunteer; Experimental 2-ICD; Experimental 3-Healthy volunteer; Experimental 3-ICD
Drug: Oral RJ026 capsules — Both the oral dosage form and the inhalation solution share the identical active ingredient.
  Arms: Active Comparator-Healthy volunteer; Active Comparator-ICD

SUMMARY:
This Phase 1 clinical trial investigates the pharmacokinetics and safety profile of single-dose inhaled RJ026 in healthy volunteers and patients with interstitial lung disease (ILD). The randomized, double-blind, dose-escalation study employs a parallel-group design with three inhaled dose cohorts (4mg, 8mg, and 12mg) and one oral comparator arm, enrolling a total of 42 patients (12 per inhaled group, 6 in oral group) and 42 healthy volunteers (12 per inhaled group, 6 in oral group). The trial features comprehensive pharmacokinetic sampling through 15 timed blood collections over 24 hours and bronchoalveolar lavage at specified intervals (1h, 6h, 12h, or 24h post-dose) to characterize both systemic and pulmonary drug exposure. The study incorporates rigorous safety monitoring including adverse event tracking, vital sign measurements, and laboratory assessments over a 7-day observation period following drug administration. Conducted at Shanghai Jiao Tong University's Ruijin Hospital over a 12-month period (July 2025-July 2026), this investigation aims to establish the foundational pharmacokinetic parameters and safety profile of RJ026 delivery in ILD patients while comparing pulmonary bioavailability against conventional oral administration.

ELIGIBILITY:
ICD patients:

Inclusion Criteria:

1. Age ≥40 years, any gender
2. Diagnosed or suspected ILD (IPF or CTD-ILD) based on HRCT or thin-section CT
3. FVC ≥40% predicted, DLCO ≥40% predicted, FEV1/FVC ≥0.7
4. Able to tolerate bronchoscopy
5. Willing to use effective contraception during study
6. Capable of proper inhaler use

Exclusion Criteria:

1. Pregnancy or lactation
2. Allergy to study drug components
3. Active respiratory infection or acute cardiopulmonary disease
4. Abnormal liver function (ALT/AST/GGT > ULN or total bilirubin > ULN)
5. Recent smoking (within 6 months) or alcohol abuse
6. Participation in other clinical trials within 3 months
7. Blood donation ≥400mL within 3 months
8. HBV DNA ≥2000 IU/mL or HCV RNA ≥1000 IU/mL or HIV positive

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
AUC0-24 hours of blood samples in ILD patients | Baseline, 10 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose
  AUC0-24 hours: Area Under the plasma concentration-time Curve from time zero to 24 hours post dose. Plasma pharmacokinetic (PK) parameters of RJ026 in ILD patients.

SECONDARY OUTCOMES:
AUC0-∞ of blood samples in ILD patients | Baseline, 10 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose
  AUC0-∞: Area Under the plasma concentration-time Curve from time zero to infinity. Plasma pharmacokinetic (PK) parameters of RJ026 in ILD patients.
Tmax of blood samples in ILD patients | Baseline, 10 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose
  Tmax: Time to reach maximum plasma concentration. Plasma pharmacokinetic (PK) parameters of RJ026 in ILD patients.
Cmax of blood samples in ILD patients | Baseline, 10 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose
  Cmax: Peak Plasma Concentration. Plasma pharmacokinetic (PK) parameters of RJ026 in ILD patients.
T1/2 of blood samples in ILD patients | Baseline, 10 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose
  T1/2: Half-life. Plasma pharmacokinetic (PK) parameters of RJ026 in ILD patients.
AUC0-24 hours of BALF (Bronchoalveolar Lavage Fluid) samples in ILD patients | 1 hours, 6 hours, 12 hours, and 24 hours post-dose
  AUC0-24 hours: Area Under the BALF concentration-time Curve from time zero to 24 hours post-dose. Lung pharmacokinetic (PK) parameters of RJ026 in ILD patients.
AUC0-∞ of BALF (Bronchoalveolar Lavage Fluid) samples in ILD patients | 1 hours, 6 hours, 12 hours, and 24 hours post-dose
  AUC0-∞: Area Under the BALF concentration-time Curve from time zero to infinity. Lung pharmacokinetic (PK) parameters of RJ026 in ILD patients.
Tmax of BALF (Bronchoalveolar Lavage Fluid) samples in ILD patients | 1 hours, 6 hours, 12 hours, and 24 hours post-dose
  Tmax: Time to reach maximum BALF concentration. Lung pharmacokinetic (PK) parameters of RJ026 in ILD patients.
Cmax of BALF (Bronchoalveolar Lavage Fluid) samples in ILD patients | 1 hours, 6 hours, 12 hours, and 24 hours post-dose
  Cmax: Peak BALF Concentration. Lung pharmacokinetic (PK) parameters of RJ026 in ILD patients.
T1/2 of BALF (Bronchoalveolar Lavage Fluid) samples in ILD patients | 1 hours, 6 hours, 12 hours, and 24 hours post-dose
  T1/2: Half-life. Lung pharmacokinetic (PK) parameters of RJ026 in ILD patients.
AUC0-24 hours of blood samples in healthy volunteers | Baseline, 10 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose
  AUC0-24 hours: Area Under the plasma concentration-time Curve from time zero to 24 hours post-dose. Lung pharmacokinetic (PK) parameters of RJ026 in healthy volunteers
AUC0-∞ of blood samples in healthy volunteers | Baseline, 10 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose
  AUC0-∞: Area Under the plasma concentration-time Curve from time zero to infinity. Plasma pharmacokinetic (PK) parameters of RJ026 in healthy volunteers.
Tmax of blood samples in healthy volunteers | Baseline, 10 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose
  Tmax: Time to reach maximum plasma concentration. Plasma pharmacokinetic (PK) parameters of RJ026 in healthy volunteers.
Cmax of blood samples in healthy volunteers | Baseline, 10 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose
  Cmax: Peak Plasma Concentration. Plasma pharmacokinetic (PK) parameters of RJ026 in healthy volunteers.
T1/2 of blood samples in healthy volunteers | Baseline, 10 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, and 24 hours post-dose
  T1/2: Half-life. Plasma pharmacokinetic (PK) parameters of RJ026 in healthy volunteers.
Incidence of adverse events and serious adverse events. | Through study completion, an average of 7 days
  Safety Evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No